CLINICAL TRIAL: NCT07229755
Title: Comparison Between Effect of Empirical Antibiotic Prophylaxis Versus Enhanced Prophylactic Measures on Rate of Urinary Tract Infection After Flexible Ureteroscopy in Children With Pyuria
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU MS591/2024
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Urinary Tract Infection (Diagnosis)
MeSH Terms: conditions — Urinary Tract Infections; Disease | interventions — Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- empirical antibiotic prophylaxis (Placebo Comparator): empirical antibiotic not culture guided
  Interventions: Drug: Ceftriaxone (Rocephin®); Device: Levofloxacin
- enhanced antibiotic prophylaxis (Experimental)
  Interventions: Drug: Ceftriaxone (Rocephin®); Device: Levofloxacin

INTERVENTIONS:
Drug: Ceftriaxone (Rocephin®) — empirical antibiotic vs urine culture guided antibiotic
Device: Levofloxacin — culture based antibiotic

SUMMARY:
The aim of this study is to compare between effect of empirical antibiotic prophylaxis versus enhanced prophylactic measures on rate of urinary tract infection after Flexible ureteroscopy in Children.

ELIGIBILITY:
Inclusion Criteria:

* Age starting from 4 up to 14 years old.
* Patients with renal stones from 1cm to 1.5cm in largest dimensions (not more than 4 cm3 measured by CTUT) undergoing flexible URS.

Exclusion Criteria:

* Patients who refuse to participate in the study.
* Patients with single functioning kidney.
* Patients with rising serum creatinine.
* Known patient with neurogenic bladder.
* Patients with DM type1.
* Immunocompromised children.

  * Children with coagulopathy.
  * Patients with untreated UTI (or any interfering symptoms with UTI as fever or irritative LUTS).

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Decreased rate of urinary tract infection after Flexible ureteroscopy in Children | From enrollment to the end of treatment at 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diaa El din Mahmoud, Proffessor, Study Director — Ain Shams University; Mohamed Saied, Lecturer, Study Director — Ain Shams University; Hisham Arafa, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Akram M, Jahrreiss V, Skolarikos A, Geraghty R, Tzelves L, Emilliani E, Davis NF, Somani BK. Urological Guidelines for Kidney Stones: Overview and Comprehensive Update. J Clin Med. 2024 Feb 16;13(4):1114. doi: 10.3390/jcm13041114. PMID 38398427